CLINICAL TRIAL: NCT03163537
Title: Disturbing Factors and Stress Levels in Vascular Surgeons During Kidney Transplantations
Brief Title: Disturbing Factors in the Operating Room
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HEEL-2016-01
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Disturbing Factors; Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Kidney transplantation, postmortal, day
  Interventions: Device: HealthPatch
- Kidney transplantation, postmortal, night
  Interventions: Device: HealthPatch
- Kidney transplantation, living donor
  Interventions: Device: HealthPatch

INTERVENTIONS:
Device: HealthPatch — Smart patch that is able to measure stress real time using an algorithm between HR and HRV

SUMMARY:
Observation of disturbing factors in the operating room and comparison between day and night shift. The investigators have chosen to observe kidney transplantations, since this type of operation has the same priority during day and night. Stress levels of surgeons will be measured using the HealthPatch.

ELIGIBILITY:
Inclusion Criteria:

* All vascular surgeons who are able to perform elective as well as postmoral kidney transplantations

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Vascular surgeons during kidney transplantation
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-13 (Actual)

PRIMARY OUTCOMES:
Factors that are disturbing for vascular surgeons during kidney transplantations | 2 hours
  One investigator will report all factors that potentially disturb the vascular surgeon during kidney transplantation. Nature and severity of the disturbing factors will be reported, such as opening and closing of doors, beepers. For this, the investigators will use an observational tool for assessing surgical flow disruptions (Parker SE, et al. Development and evaluation of an observational tool for assessing surgical flow disruptions and their impact on surgical performance. World J Surg 2010; 34(2): 353-361)

SECONDARY OUTCOMES:
Stress levels | 2 hours
  Stress levels, measured by the HealthPatch
State Trait Anxiety Inventory | 5 minutes
  STAI; anxiety questionnaire